CLINICAL TRIAL: NCT04938141
Title: Medical Events of Interest and Health-Related Quality of Life in Chronic Lymphocytic Leukemia Patients Initiating Treatment With Bruton's Tyrosine Kinase Inhibitors Acalabrutinib or Ibrutinib
Brief Title: MEOI and HRQoL in CLL Patients Treated With BTKis
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8220R00036
Record Dates: First submitted 2021-06-17; First posted 2021-06-24 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-04

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Acalabrutinib: CLL patients initiating acalabrutinib alone or in combination with an anti-CD20 mAb
- Ibrutinib: CLL patients receiving ibrutinib alone or in combination with an anti-CD20 mAb

SUMMARY:
This is a multi-site observational study of medical events of interest (MEOI) and health-related quality of life (HRQoL) in chronic lymphocytic leukemia (CLL) patients initiating treatment with the Bruton's tyrosine kinase inhibitors (BTKi) acalabrutinib or ibrutinib in the United States (US)

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Physician-confirmed diagnosis of CLL or small lymphocytic lymphoma (SLL)
* BTKi naïve patients who initiate acalabrutinib or ibrutinib treatment alone or in combination with an anti-CD20 mAb within 7 days (before or after) study enrollment*. Both treatment naïve and relapsed/refractory CLL patients will be included.
* Provides informed consent
* Adequate English reading skills
* Able to access and use a computer, tablet, or smartphone to complete PROs

Exclusion Criteria:

* Use of BTKi any time prior to study enrollment.
* Currently receiving systemic treatment for another malignancy
* Currently enrolled in a clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients who have recently initiated treatment for CLL/SLL with acalabrutinib or ibrutinib in the front-line or relapsed/refractory setting
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Patient Characteristics | Baseline
  To describe the demographic and clinical characteristics of CLL patients who have recently initiated acalabrutinib or ibrutinib.
Chart Recorded Medical Events of Interest | 24 Month Follow-up
  To describe MEOI experienced by CLL patients who have recently initiated acalabrutinib or ibrutinib using medical chart abstracted data, over a 24-month period
Patient Reported Medical Events of Interest | 24 month follow-up
  To describe MEOI experienced by CLL patients who have recently initiated acalabrutinib or ibrutinib using patient reported data, over a 24-month period.
HRQoL | 24 month follow-up
  To describe HRQoL for CLL patients who recently initiated acalabrutinib or ibrutinib using patient reported data, over a 24-month period

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Research Site, Fountain Valley, California
  - Research Site, Redlands, California
  - Research Site, Boca Raton, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Savannah, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Jackson, Mississippi
  - Research Site, Berkeley Heights, New Jersey
  - Research Site, Amherst, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, York, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/